CLINICAL TRIAL: NCT02422888
Title: Reducing Micro Vascular Dysfunction In Revascularized ST-elevation Myocardial Infarction Patients by Off-target Properties of Ticagrelor
Brief Title: Reducing Micro Vascular Dysfunction in Acute Myocardial Infarction by Ticagrelor
Acronym: REDUCE-MVI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Erasmus Medical Center (Other); Hospital San Carlos, Madrid (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Maarten van Leeuwen, Study coordinator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10048; 2014-005363-33 (EudraCT Number)
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Myocardial Infarction
Keywords: ST elevation myocardial infarction; Percutaneous coronary intervention; Endothelial function; Ticagrelor; Prasugrel
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90 mg twice a day, tablet Duration: 1 year after PCI
  Interventions: Drug: Ticagrelor
- Prasugrel (Active Comparator): Prasugrel 10 mg once a day, tablet Duration: 1 year after PCI
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor — After a standard loading dose of 180 mg ticagrelor in the ambulance (before primary PCI), patients will receive a maintenance dose of ticagrelor 90 mg twice a day for 1 year.
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Prasugrel — After a standard loading dose of 180 mg ticagrelor in the ambulance (before primary PCI), patients will receive a single loading dose of prasugrel 60 mg (1 day after standard loading dose ticagrelor),followed by a maintenance dose of prasugrel 10 mg once a day for 1 year.
  Other Names: Efient
  Arms: Prasugrel

SUMMARY:
The current trial will compare the protective effect of ticagrelor and prasugrel on microvascular dysfunction in patients with revascularized ST elevation myocardial infarction.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction is highly prevalent in revascularized ST-elevation myocardial infarction and has important prognostic implications. Current data suggest that ticagrelor might be superior to prasugrel in the reduction of coronary microvasculature dysfunction. Thus, we have designed a clinical trial that will compare microvascular function in revascularized ST-elevation myocardial infarction patients at treatment steady state with ticagrelor or prasugrel. Coronary microvascular dysfunction will be assessed with the index of microcirculatory resistance after primary percutaneous coronary intervention and at 1 month follow-up in the infarct-related vessel and non-infarct related vessel.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Patients presenting with ST-elevation myocardial infarction <12 hours after symptom onset
3. Successful percutaneous coronary intervention of the infarct-related vessel with a modern drug-eluting stent
4. Intermediate stenosis in non-infarct-related vessel (50-90%)

Exclusion Criteria:

1. history of myocardial infarction
2. Participation in another clinical study with an investigational product during the preceding 30 days
3. history of cerebrovascular accident (CVA) or 'transient ischaemic attack' (TIA)
4. History of intracranial haemorrhage
5. indication or use of oral anticoagulant therapy (i.e. acenocoumarol)
6. severe liver dysfunction (Child-Pugh score 10-15)
7. congestive heart failure
8. cardiogenic shock
9. left ventricular ejection fraction < 35%
10. bleeding diathesis
11. age ≥ 75 or < 18
12. body weight < 60 kg
13. gout
14. coagulation disorders
15. severe pulmonary disease
16. pregnancy and breast feeding
17. limited life expectancy
18. platelet count < 100 000/mm3
19. history of drug addiction or alcohol abuse in the past 2 years
20. need for chronic nonsteroidal anti-inflammatory drug
21. creatinine clearance <30 mL/min or dialysis
22. chronic total occlusion (CTO)
23. Left main disease
24. allergy or contra-indication for ticagrelor or prasugrel
25. Contra-indication for adenosine
26. Patients unable to be followed on-site
27. Unable to undergo or contra-indications for MRI
28. Contra-indication for drug-eluting stent
29. Inability to obtain informed consent
30. Coronary artery bypass grafting in medical history

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Index of microcirculatory resistance (IMR) | 1 month after primary PCI
  measured in the infarct-related artery

SECONDARY OUTCOMES:
Delta Index of microcirculatory resistance (IMR) | Baseline vs. 1 month follow-up
  measured in the infarct-related artery and non-infarct related artery
The reactive hyperemia index (RHI) | 1 month and 1 year after primary PCI
Myocardial salvage | 1 month after primary PCI
  measured with MRI
Left ventricular ejection fraction (LVEF) recovery | 1 month after primary PCI
  measured with MRI
Microvascular obstruction | 3 days after primary PCI
  measured with MRI
Asymmetric Dimethylarginine (ADMA) levels | 1 month after primary PCI
  Blood measurements
Intra-myocardial haemorrhage | 3 days after primary PCI
  measured with MRI

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Wang L, Travieso A, van der Hoeven N, van Leeuwen MAH, Janssens G, Mejia-Renteria H, Jeronimo A, Gonzalo N, Nijveldt R, van Royen N, Escaned J. Improved Nonculprit Stenosis Assessment in Patients With ST-Segment Elevation Myocardial Infarction Using Quantitative Flow Ratio. JACC Cardiovasc Interv. 2023 Jul 24;16(14):1828-1830. doi: 10.1016/j.jcin.2023.04.045. Epub 2023 May 19. No abstract available. PMID 37204397
- [Derived] van der Hoeven NW, Janssens GN, Everaars H, Nap A, Lemkes JS, de Waard GA, van de Ven PM, van Rossum AC, Escaned J, Mejia-Renteria H, Ten Cate TJF, Piek JJ, von Birgelen C, Valgimigli M, Diletti R, Riksen NP, Van Mieghem NM, Nijveldt R, van Leeuwen MAH, van Royen N. Platelet Inhibition, Endothelial Function, and Clinical Outcome in Patients Presenting With ST-Segment-Elevation Myocardial Infarction Randomized to Ticagrelor Versus Prasugrel Maintenance Therapy: Long-Term Follow-Up of the REDUCE-MVI Trial. J Am Heart Assoc. 2020 Mar 3;9(5):e014411. doi: 10.1161/JAHA.119.014411. Epub 2020 Mar 3. PMID 32122216
- [Derived] van Leeuwen MAH, van der Hoeven NW, Janssens GN, Everaars H, Nap A, Lemkes JS, de Waard GA, van de Ven PM, van Rossum AC, Ten Cate TJF, Piek JJ, von Birgelen C, Escaned J, Valgimigli M, Diletti R, Riksen NP, van Mieghem NM, Nijveldt R, van Royen N. Evaluation of Microvascular Injury in Revascularized Patients With ST-Segment-Elevation Myocardial Infarction Treated With Ticagrelor Versus Prasugrel. Circulation. 2019 Jan 29;139(5):636-646. doi: 10.1161/CIRCULATIONAHA.118.035931. PMID 30586720
- [Derived] Janssens GN, van Leeuwen MAH, van der Hoeven NW, de Waard GA, Nijveldt R, Diletti R, Zijlstra F, von Birgelen C, Escaned J, Valgimigli M, van Royen N. Reducing Microvascular Dysfunction in Revascularized Patients with ST-Elevation Myocardial Infarction by Off-Target Properties of Ticagrelor versus Prasugrel. Rationale and Design of the REDUCE-MVI Study. J Cardiovasc Transl Res. 2016 Jun;9(3):249-256. doi: 10.1007/s12265-016-9691-3. Epub 2016 Apr 21. PMID 27102290